CLINICAL TRIAL: NCT04257474
Title: Barriers to Screening Breast MRI Utilization Among Patients at Elevated Risk (B-SUPER)
Brief Title: Barriers to Screening Breast MRI Utilization Among Patients at Elevated Risk
Acronym: B-SUPER
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-20257
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Pathogenic BRCA 1/2 Mutation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assessing Health Services Utilization Model (HSUM): 150 women with a high lifetime breast cancer risk will be recruited from mammography and primary care clinics. Researchers will assess HSUM factors influencing screening breast MRI utilization. Results will identify participant-level HSUM factors significantly associated with screening outcomes.
  Interventions: Behavioral: Self-Report Survey
- Qualitative Interviews: Researchers will randomly select 30 participants from group 1 and will use semi-structured qualitive interviews exploring factors impacting utilization of screening breast MRI
  Interventions: Behavioral: Qualitative Interviews

INTERVENTIONS:
Behavioral: Self-Report Survey — The self-report survey will be created using the Health Services Utilization Model (HSUM)
  Groups: Assessing Health Services Utilization Model (HSUM)
Behavioral: Qualitative Interviews — Researchers will randomly select 30 participants from group 1 and will use semi structured qualitive interviews exploring factors impacting utilization of screening breast MRI
  Groups: Qualitative Interviews

SUMMARY:
This study seeks to develop an explanatory framework for breast MRI utilization to inform future interventions. The Health Services Utilization Model (HSUM) will guide the selection of specific participant-level factors for examination, including predisposing characteristics (knowledge, health/cultural beliefs), enabling resources (social support, cost/insurance coverage), and perceived need (perceived susceptibility, provider recommendation).

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak/read English
* Within 2 years of last screening mammogram
* Pathogenic BRCA1/2 mutations OR estimated lifetime risk ≥20% per the National Cancer Institute (NCI) Breast Cancer Risk Assessment Tool (BCRAT)

Exclusion Criteria:

* Women who have received a prior diagnosis of breast cancer

Ages: 25 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — The lifetime risk for breast cancer in men is very low (1.2% for male BRCA1 mutation carriers and 6.8% for male BRCA2 mutation carriers).
Study Population: Women will be recruited from mammography and primary care clinics, community-based outreach events, or via Facebook
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vadaparampil, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Self-Report Surveys Only: Women with a high lifetime breast cancer risk were recruited from mammography and primary care clinics. Group 1 took a self-report survey that was created using the Health Services Utilization Model (HSUM)
- Group 2:Self-Report Survey and Qualitative Interviews: Women with a high lifetime breast cancer risk were recruited from mammography and primary care clinics.
  Self-Report Survey: The self-report survey was created using the Health Services Utilization Model (HSUM)
  Researchers randomly selected participants from group 1 who took self-report Survey and held semi-structured qualitive interviews exploring factors impacting utilization of screening breast MRI
Period: Overall Study
Arm/Group | Group 1: Self-Report Surveys Only | Group 2:Self-Report Survey and Qualitative Interviews
Started | 172 | 63
Completed | 172 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Self-Report Survey and Qualitative Interviews: Women with a high lifetime breast cancer risk were recruited from mammography and primary care clinics.
  Self-Report Survey: The self-report survey was created using the Health Services Utilization Model (HSUM)
  Researchers randomly selected participants from group 1 who took self-report Survey and held semi-structured qualitive interviews exploring factors impacting utilization of screening breast MRI
- Total: Total of all reporting groups
Arm/Group | Group 1: Self-Report Surveys Only | Group 2: Self-Report Survey and Qualitative Interviews | Total
Number analyzed (Participants) | 172 | 63 | 235
Age, Customized [Count of Participants; unit: Participants]
  25-29 | 20 | 3 | 23
  30-39 | 62 | 18 | 80
  40-49 | 38 | 12 | 50
  50-59 | 28 | 19 | 47
  60-69 | 17 | 10 | 27
  70-79 | 5 | 1 | 6
  80-85 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 63 | 235
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 164 | 60 | 224
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 149 | 54 | 203
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 8 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 172 | 63 | 235

OUTCOME MEASURES:

1. Primary Outcome: Reporting Receipt of MRI Breast Screening at Any Time
Description: Participant-reported receipt of screening breast MRI at any time in the past.
Time Frame: Baseline
Population: This study uses a mixed-methods design. All data from participants who completed self-report surveys were analyzed as one group. Semi-structured interviews were done to understand more about the patients decisions, not to compare any group against another.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: All participants who completed self-report surveys in addition to participants who completed self-report surveys and also completed semi structured interviews.
Arm/Group | All Participants
Number analyzed (Participants) | 235
percentage of participants | 32.34

2. Primary Outcome: Reporting Receipt of MRI Breast Screening in the Last 24 Months
Description: Participant-reported receipt of screening breast MRI in the last 24 months
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 235
percentage of participants | 25.11

3. Secondary Outcome: Reporting Receipt of Mammogram
Description: Participant-reported receipt of breast cancer screening mammogram in the last 24 months
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 235
percentage of participants | 71.06

4. Secondary Outcome: Reporting Receipt of Ultrasound
Description: Participant-reported receipt of breast cancer screening ultrasound in the last 24 months
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 235
percentage of participants | 34.04

5. Secondary Outcome: Reporting Receipt of Chemoprevention
Description: Participant-reported receipt of chemoprevention at any point in time (including currently receiving).
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 235
percentage of participants | 18.30

6. Secondary Outcome: Reporting Receipt of Genetic Testing
Description: Participant-reported receipt of genetic testing at any time in the past
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 235
percentage of participants | 42.99

7. Secondary Outcome: Reporting Receipt of Genetic Counseling
Description: Participant-reported receipt of genetic counseling at any time in the past
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 235
percentage of participants | 39.57

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected for this project.
Description: Adverse Events were not collected for this project.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT04257474/Prot_SAP_000.pdf